CLINICAL TRIAL: NCT02320331
Title: Partnerships to Improve Lifestyle Interventions (PILI) 'Ohana Dissemination Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Kula No Na Po'e Hawaii (Other); Ke Ola Mamo (Other); Hawai'i Maoli (Other); Kokua Kalihi Valley (Unknown)
Responsible Party: Principal Investigator, Joseph Keawe'aimoku Kaholokula, Professor and Chair, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD001660
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (1):
- PILI Lifestyle Program (Experimental)
  Interventions: Behavioral: PILI Lifestyle Program

INTERVENTIONS:
Behavioral: PILI Lifestyle Program — A 12-week Individual-focused Behavioral Weight Loss Intervention. Our 12-week intervention is modeled after the Diabetes Prevention Program's (DPP) Lifestyle Intervention. Each of the 8 lessons of this 12-week intervention will be done in a group classroom setting via trained community peer educators for a total of 8 group meetings as outlined above. Lesson 1 through 4 will be done every week, once a week, for 4 weeks followed by every other week for the remaining 4 lessons (lessons 5 through 8). Each group meeting will have between 12 to 15 people and take 1 to 1 ½ hours to complete. After completing the 12-week behavioral weight loss intervention, participants will participate in an additional 6 lessons. A lesson will be done once-a-month. These 6 lessons will teach participants how to involve their family and friends in their healthy lifestyle changes.

SUMMARY:
The purpose of the OHA PILI 'Ohana Project is to disseminate and evaluate the effectiveness of a community-based intervention (PILI 'Ohana Intervention Program) aimed at eliminating obesity in Pacific Peoples across the four islands. Dissemination will involve implementation of the program in eight communities through partnerships with nine different community-based organizations serving those areas (four founding community partners and five new community partners). These organizations provide services to a large number of Pacific Peoples, including (but not limited to) Native Hawaiians, Samoans, Filipinos, and Chuukese.

The main aims are to: (1) train five additional community organizations and their staff to deliver the PILI 'Ohana Intervention Program, (2) to enroll 150 overweight/obese participants across 8 different communities and four different islands into the intervention program, and (3) to evaluate the effectiveness of the program in reducing weight/BMI by at least 3% of the participant's initial weight.

The PILI 'Ohana Intervention is a 9-month lifestyle intervention focusing on individual health behaviors in the context of family and community environments and in the socio-cultural context of Pacific Peoples. In order to increase the likelihood that an organization will implement the PLP, they will be able to adapt the intervention and participant assessments. The POP will provide guidance on adaption of the intervention and assessments at the training (CHS #21680). What is described below is the maximum amount of contact and assessment procedures that participants will undergo. Therefore, organizations may change the timing of the 14 lessons and refrain from using all the assessment procedures, but will still provide the 14 lessons and offer the same incentives to participants for assessments.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 25
* Clients and/or residents of communities served by 9 partnering community organizations

Exclusion Criteria:

-

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 9 months
  Weight at 9 months compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Native Hawaiian Health, University of Hawaii, Honolulu, Hawaii, United States